CLINICAL TRIAL: NCT01412671
Title: Special Drug Use Investigation of Nexavar (Unresectable or Advanced Renal Cell Carcinoma: Early Access Program)
Brief Title: Nexavar Post-marketing Surveillance for RCC in Japan: Early Access Program
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15037; NEXAVAR-RCC-01 (Other: Company Internal)
Record Dates: First submitted 2011-08-07; First posted 2011-08-09 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Carcinoma, Renal Cell
Keywords: Nexavar; unresectable or advanced renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Patients who have received Nexavar for unresectable or advanced RCC.

SUMMARY:
This study is an early access program of 'Nexavar post-marketing surveillance (PMS) for renal cell carcinoma (RCC) in Japan' which is a regulatory, local prospective and observational study for patients with unresectable or advanced RCC under real-life practice conditions. The objective of this study is to assess safety and effectiveness of Nexavar at some limited sites which joined to clinical trial of Nexavar, before available of it in the market. The enrollment period is 2 months, and patients who received Nexavar will be recruited and followed one year since starting Nexavar administration. The data of this study will be integrated into the Nexavar PMS and the data will not be analyzed and reported alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received Nexavar for unresectable or advanced renal cell carcinoma

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is patients who received Nexavar for unresectable or advanced RCC.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2008-02-27 (Actual); Primary Completion 2011-09-21 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions and serious adverse events in subjects who received Nexavar | After Nexavar administration, up to 1 year

SECONDARY OUTCOMES:
Incidence of adverse drug reactions in subpopulation in a variety of baseline data [such as demographic data, concomitant disease, clinical staging of RCC, Eastern Cooperative Oncology Group-Performance Status (ECOG-PS)] | After Nexavar administration, up to 1 year
Effectiveness evaluation assessment [overall survival, response rate, stable disease rate, progression disease rate] by investigator-determined overall best response [according to the General rule for clinical and pathological studies on RCC] | After Nexavar administration, up to 1 year
The status of therapy with Nexavar [duration of treatment, daily dose] | After Nexavar administration, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan